CLINICAL TRIAL: NCT03200171
Title: Effect of Direct Acting Antiviral Agents on Behavior of Hepatocellular Carcinoma and Overall Survival in Patients With Chronic Hepatitis C
Brief Title: Effect of DAAs on Behavior of HCC in HCV Patients
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: Helwan University (Other); Cairo University (Other); Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Alboraie, Principal Investigator, Al-Azhar University
Other Study IDs: EARTH-HCC-1
Record Dates: First submitted 2017-06-24; First posted 2017-06-27 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma, Hepatocellular; Hepatitis C
Keywords: Carcinoma, Hepatocellular; Hepatitis C
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: HCC patients who received DAAs for chronic HCV previously (either responders or not)
- Group II: HCC patients who are naive to DAAs.

SUMMARY:
Investigators aim to study the effect of direct acting antiviral agents (DAAs) on behavior of hepatocellular carcinoma (HCC) and overall survival in patients with chronic hepatitis C (CHC).

DETAILED DESCRIPTION:
Introduction:

Chronic hepatitis C (HCV) infection can be complicated with liver cirrhosis and subsequently hepatocellular carcinoma (HCC). HCC develops at an annual rate of 1% to 4%, although higher rates up to 7% have been reported in Japan. Recently; Reig et al; noticed that there was an unexpected high rate of early tumor recurrence in patients with HCV-related HCC undergoing interferon-free therapy (1). After this report; many publications have discussed the issue of HCC development and recurrence in HCV patients treated with interferon free regimens. Results of these trials are controversial with no definite conclusion till today. There is an unmet need for further study the effect of interferon free regimens on development of de novo HCC, recurrence of HCC and behavior of HCC in chronic HCV patients.

Aim of the study:

Investigators aim to study the effect of direct acting antiviral agents (DAAs) on behavior of hepatocellular carcinoma (HCC) and overall survival in patients with chronic hepatitis C (CHC).

Materials & methods:

Study Design: Prospective case control study

* Setting: Multicenter study
* Patients: 300 patients will be recruited in 2 groups assignment .
* Methods:

Procedure of data collection

The following data will be collected at base line for each patient:

1. Medical history: including current and previous treatment with stress on History of treatment by DAAs (date started, used regimen, duration of treatment and treatment response)
2. Full clinical examination
3. Laboratory Investigations:

   1. Complete blood picture (CBC):
   2. Liver profile: alanine aminotransferase (ALT), aspartate aminotransferase (AST), albumin, total and direct bilirubin, prothrombin time and international normalized ratio.
   3. Renal profile: serum blood urea nitrogen (BUN), creatinine, sodium and potassium levels.
   4. Hepatitis markers: hepatitis B surface antigen (HBs Ag) and hepatitis C virus antibody (HCV Ab).
   5. Alpha feto protein (AFP)
   6. Tri-Phasic spiral abdominal CT: to diagnose HCC by typical vascular pattern and to assess tumor extension.
   7. Biopsy if needed After confirming HCC diagnosis, included patients will be classified according to barcelona clinic liver cancer (BCLC) staging system and standard of care treatment will be provided to patients with different stages according to BCLC guidelines.

Follow up schedule:

Patients will be followed by CT scan or MRI examination and routine liver tests including AFP every 3 months during the first 2 years then every 6 months during the subsequent 3 years if no evidence of HCC recurrence during the first 2 years' period (for all patients regardless HCC treatment receipt and its type). Local recurrence will be defined as reappearance of tumor adjacent to the treated site of the initial HCC and distant recurrence as the emergence of one or several tumor(s) not adjacent to the treated zone. Criteria for the diagnosis of HCC recurrence will be the same as initial HCC, i.e. presence of typical hallmark of HCC according to European Association for the Study of the Liver - European Organisation for Research and Treatment of Cancer (EASL-EORTC) guidelines and defined by presence on imaging of hyper vascular in the arterial phase with washout in the portal venous or delayed phases. All imaging exams will be centralized and assessed by the same radiologist.

Analysis of results:

- Statistical analysis will aim at identifying factors leading to change of behavior of HCC after DAAs in CHC patients in addition to determination of the overall survival in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCV related Hepatocellular carcinoma (HCC); all patients with confirmed diagnosis of HCC according to EASL-EORTC guidelines who attend HCC outpatient clinics in the study centers will be enrolled after signing informed consent. Patients will be then assigned into two main comparison groups:
* Group I: HCC patients who received DAAs for chronic HCV previously (either responders or not)
* Group II: HCC patients who are naive to DAAs.

Exclusion Criteria:

* Patients who refuse to be enrolled in the study.
* Patients with hepatitis B virus or any other causes of cirrhosis.
* Other prior malignancy without complete remission in the last five years, with the exception of adequately treated basal cell carcinoma or in situ cervical cancer; in case of other prior malignancy, the diagnosis of HCC has to be histologically proven.
* HCC developed on transplanted liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCV related Hepatocellular carcinoma (HCC)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 6 months - 3 years
  he length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Behavior of hepatocellular carcinoma | 6 months - 3 years
  Early recurrence, or rapid progression

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 6 months - 3 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. Progression-free survival (PFS) will be measured by the Independent Radiological Review according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alboraie, M.D., Principal Investigator — Al-Azhar University
Locations (3):
- Egypt (3):
  - MOHAMED Alboraie, Cairo
  - Helwan University, Cairo
  - National Hepatology and Tropical Medicine Research Institute, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reig M, Marino Z, Perello C, Inarrairaegui M, Ribeiro A, Lens S, Diaz A, Vilana R, Darnell A, Varela M, Sangro B, Calleja JL, Forns X, Bruix J. Unexpected high rate of early tumor recurrence in patients with HCV-related HCC undergoing interferon-free therapy. J Hepatol. 2016 Oct;65(4):719-726. doi: 10.1016/j.jhep.2016.04.008. Epub 2016 Apr 13. PMID 27084592